CLINICAL TRIAL: NCT04160169
Title: Counseling on Injectable Contraception and HIV Risk: Evaluation of a Pilot Intervention in Tanzania
Brief Title: Counseling on Injectable Contraception and HIV Risk in Tanzania
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Ministry of Health, Tanzania (Other Government); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Other Study IDs: 18-1049
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Contraception
Keywords: Counseling; Tanzania

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Counseling messages on injectable use and HIV acquisition risk — Counseling messages based on 2017 World Health Organization guidance, a review of the Strategic Communication Framework for Hormonal Contraceptive Methods and Potential HIV-related Risks, and the Family Planning Global Handbook were provided to clients expressing interest in injectables during regular family planning appointments.

SUMMARY:
The main objective of the evaluation was to assess the effect of providing injectable and HIV risk counseling messages on contraceptive knowledge and behavior during a three month pilot intervention in ten healthcare facilities in Tanzania.

DETAILED DESCRIPTION:
The evaluation assessed the effect of providing injectable and HIV risk counseling messages on contraceptive knowledge and uptake during a three month pilot intervention. The intervention was conducted September-November 2018 in ten healthcare facilities located in the Iringa and Njombe regions of Tanzania. Data collection for the evaluation occurred November-December 2018 and included 471 client exit interviews, 26 healthcare provider interviews, and the extraction of monthly aggregate service statistics for 12 months prior to the intervention and three months of the intervention. Univariate and bivariate analyses were used to assess quantitative interview data. Thematic qualitative assessment was used to assess qualitative interview data from healthcare providers. Interrupted time series analysis was used to assess changes in the trend of monthly contraceptive uptake.

ELIGIBILITY:
Inclusion Criteria:

* Expressed interest in injectable use
* HIV-negative or unknown HIV status

Exclusion Criteria:

* Positive HIV status known to healthcare provider

Ages: 15 Years to 49 Years | Sex: Female
Age Groups: Child, Adult
Study Population: All women attending a participating healthcare facility during the three month intervention period and who met eligibility criteria received the hormonal contraception and HIV risk messages.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Number of clients obtaining an injectable during their family planning appointment | After implementation of counseling messages, up to 13 weeks
  Injectable uptake of interviewed clients
Percent of clients obtaining an injectable during their family planning appointment | After implementation of counseling messages, up to 13 weeks
  Injectable uptake of interviewed clients
Monthly total number of family planning clients by method obtained | September 2017 through November 2018
  Contraceptive uptake during pilot intervention

SECONDARY OUTCOMES:
Number of correct hormonal contraception and HIV risk counseling messages mentioned during spontaneous recall | After implementation of counseling messages, up to 13 weeks
  Knowledge of hormonal contraception and HIV risk messages
Percent of correct hormonal contraception and HIV risk counseling messages mentioned during spontaneous recall | After implementation of counseling messages, up to 13 weeks
  Knowledge of hormonal contraception and HIV risk messages
Number of correct True/False statements on hormonal contraception and HIV (11 total) | After implementation of counseling messages, up to 13 weeks
  Knowledge of hormonal contraception and HIV risk messages
Percent of correct True/False statements on hormonal contraception and HIV (11 total) | After implementation of counseling messages, up to 13 weeks
  Knowledge of hormonal contraception and HIV risk messages
Number of interviewed clients reporting an intention to use condoms as a dual method | After implementation of counseling messages, up to 13 weeks
  Intention to use condoms as a dual method
Percent of interviewed clients reporting an intention to use condoms as a dual method | After implementation of counseling messages, up to 13 weeks
  Intention to use condoms as a dual method

CONTACTS AND LOCATIONS:
Overall Officials: Janine Barden-O'Fallon, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (10):
- Tanzania (10):
  - Ilula Hospital, Ilula, Iringa
  - Mafinga Hospital, Mafinga, Iringa
  - Ihongole Health Center, Iringa
  - Ipogolo Health Center, Iringa
  - Kimande Health Center, Iringa
  - Ipelele Health Center, Njombe
  - Kibena Regional Referral Hospital, Njombe
  - Makambako Hospital, Njombe
  - Makete Hospital, Njombe
  - Njombe Health Center, Njombe

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data from the client interviews are publicly available through MEASURE Evaluation Dataverse in STATA format. The study report is also available on Dataverse.
Supporting Information: CSR
Time Frame: Data are currently available and will remain on Dataverse.org
Access Criteria: Site registration required.
URL: https://dataverse.unc.edu/dataset.xhtml?persistentId=doi:10.15139/S3/XEXQXO

REFERENCES:
- See also: Hormonal contraceptive eligibility for women at high risk of HIV: Guidance statement. 2017 — http://apps.who.int/iris/bitstream/handle/10665/254662/WHO-RHR-17.04-eng.pdf;jsessionid=035D4751CFD8B1A20F3DF079DD896C81?sequence=1
- See also: Strategic communication framework for hormonal contraceptive methods and potential HIV-related risks. 2017. — http://healthcommcapacity.org/hc3resources/strategic-communication-framework-for-hormonal-contraceptive-methods-and-potential-hiv-related-risks/
- Available data/document: Individual Participant Data Set: doi:10.15139/S3/XEXQXO — https://dataverse.unc.edu/dataset.xhtml?persistentId=doi:10.15139/S3/XEXQXO